CLINICAL TRIAL: NCT03066947
Title: A Phase I/IIa Study of SV-BR-1-GM in Metastatic or Locally Recurrent Breast Cancer Patients
Brief Title: SV-BR-1-GM in Metastatic or Locally Recurrent Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BriaCell Therapeutics Corporation (Industry)
Collaborators: Cancer Insight, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001; WRI-GEV-007 (Other: BriaCell)
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2019-12

CONDITIONS: Breastcancer; Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SV-BR-1-GM Monotherapy (Experimental): Pretreatment with low dose cyclophosphamide 2-3 days prior to SV-BR-1-GM inoculation; SV-BR-1-GM inoculation intradermally in 4 sites on the upper back (x2) and thighs (x2); Post-inoculation low dose Interferon-alpha-2b into the vaccination sites ~2 and ~4 days after SV-BR-1-GM inoculation
  Interventions: Biological: SV-BR-1-GM; Drug: Cyclophosphamide; Biological: Interferon-alpha-2b

INTERVENTIONS:
Biological: SV-BR-1-GM — See above
Drug: Cyclophosphamide — Low dose pre-treatment to reduce regulatory T cells
  Other Names: Cytoxan
Biological: Interferon-alpha-2b — Low dose given in the vaccine site to boost the immune response
  Other Names: Intron A

SUMMARY:
This is a single arm, open label study of SV-BR-1-GM, a targeted immunotherapy for breast cancer. Eligible patients will have histological confirmation of breast cancer with recurrent and/or metastatic lesions. The treatment regimen includes a pre-treatment with low-dose cyclophosphamide 2-3 days before the inoculation; inoculation in 4 sites on the thighs and upper back; and post-treatment inoculation of Interferon-alpha-2b into the sites of inoculation ~2 and ~4 days after the inoculation. These is repeated every 2 weeks for one month (3 treatments), then monthly for up to one year. Standard tumor assessments are performed at baseline and then every 2-3 months.

DETAILED DESCRIPTION:
This is a single arm, open label study of SV-BR-1-GM in recurrent and/or metastatic breast cancer. The detailed treatment regimen follows:

Pre-Inoculation Regimen:

Cyclophosphamide (Cytoxan) 300 mg/m^2 I.V., 1x only, will be given 48-72 hours before each SV-BR-1-GM inoculation, with an antiemetic of the provider's choice (steroids prohibited). If the patient is not tolerating the cyclophosphamide, a lower dose may be used (e.g. 200 or 150 mg/m^2) or it may be withheld, with the Sponsor's approval.

Innoculation Day Standard Operating Procedures:

1. Inquire regarding events of past weeks, change in medications, pain scale, ECOG scale, and review of systems.
2. Check injection sites.
3. Perform DTH skin test intra-dermally with the SV-BR-1 parent cell line (~1 x 10^6 irradiated tumor cells). Observe about 20 minutes for acute hypersensitivity. Grade III or higher acute hypersensitivity will abort therapy.
4. Inject SV-BR-1-GM intra-dermally into 4 sites in thighs and upper back (0.5 mL each). Monitor patients for 60 minutes. Vital signs will be assessed and medical attention will be warranted if unstable.

SV-BR-1-GM Preparation & Inoculation Regimen:

Each inoculation will be administered via intra-dermal injection at the investigational sites. Subjects will receive 15-25 x 10^6 viable, irradiated transfected breast tumor cells in a total volume of 2.0 ml Ringer's lactate. SV-BR-1-GM cells will be irradiated to ensure cell replication incompetency.

SV-BR-1-GM will be divided into four aliquots of 0.5 mL each and injected intra-dermally; one each into the anterior skin of the subject's right and left thighs and over the right and left upper back . Application of anesthetic lidocaine crème may be used if necessary for control of local pain before inoculation. Subjects will be monitored for 60 minutes.

After at least 10 subjects have been treated safely with this regimen, the dose of SV-BR-1-GM may be escalated or decreased in subsequent patients based on the emerging data.

Post-Inoculation Regimen:

2 days (± 1 day) after inoculation, and again 4 days (± 1 day) later after inoculation, the patient will return to the principal investigator's office to receive Interferon-alpha-2b (Merck) in 0.1 mL saline, prepared as follows: These will also be provided by the sponsor and injected intra-dermally to each inoculation site, beneath the thickest area. Again, subjects will be observed about 20 minutes. The DTH response will also be recorded at the 2 days (± 1 day) visit.

This cycle will be performed every 2 weeks for the first month of treatment (3 inoculations), and then every month for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have histological confirmation of breast cancer with recurrent and/or metastatic lesions via investigational site.

  * Patients with new or progressive breast cancer metastatic to brain will be eligible provided:

    1. There is no need for steroids and patients have not had steroids at least 2 weeks
    2. No individual tumor size is >50 mm3
    3. ECOG status <3
    4. Tumor is not impinging on Middle Cerebral Artery/speech-motor strip
    5. If surgically debulked, must be healed from surgery and at least 3 weeks have elapsed since general anesthesia
    6. Patients consent to MRI studies at 3-4 week intervals until evidence of tumor regression on at least 2 imaging studies. In no case, will the interval between MRI studies be longer than 3 months. MRI study may be introduced at any time should the patients develop new or clearly worsening symptoms and/or introduction of steroids

       2. Have evidence of persistent, recurrent, or progressive disease for which there is no known or established treatment available with curative intent, after failing at least one course of community standard systemic treatment with chemotherapy (and endocrine therapy if appropriate)

       3. Be 18 years of age or older and female

       4. Have expected survival of at least 4 months

       5. Have adequate performance status (ECOG 0-2)

       6. Patients may be maintained on hormonal therapy provided there is clear evidence of tumor progression

       7. Have provided written informed consent.

       Exclusion Criteria:

  1. Concurrent or recent chemotherapy (within 3 weeks), XRT within 3 weeks, may have had immunotherapy in the past (off within 3 weeks), or general anesthesia/major surgery (within 3 weeks). Patients must have recovered from all known or expected toxicities from previous treatment and passed a treatment-free "washout" period of 3 weeks before starting this program (8 weeks for persons receiving nitrosourea or mitomycin).
  2. History of clinical hypersensitivity to GM-CSF, Interferon-alpha-2b (Merck), yeast, beef, or to any components used in the preparation of the experimental vaccine.
  3. BUN >30 and a creatinine >2.
  4. Absolute granulocyte count < 1000; platelets <100,000.
  5. Bilirubin >2.0; alkaline phosphatase >5x upper limit of normal (ULN); ALT/AST >2x ULN.
  6. Proteinuria >1+ on urinalysis or >1 gm/24hr.
  7. Left ventricular ejection fraction (LVEF as determined by cardiac echo or MUGA scan) below the normal limits of the institutions specific testing range. This assessment may be repeated once at the discretion of the Investigator with the approval of the Sponsor.
  8. New York Heart Association stage 3 or 4 cardiac disease.
  9. A pleural effusion of moderate severity or worse.
  10. Any woman of childbearing potential, unless she:

      1. Agrees to take measures to avoid becoming pregnant during the study and
      2. Has a negative serum pregnancy test within 7 days prior to starting treatment.
  11. Women who are pregnant or nursing.
  12. Patients with concurrent second malignancy. Persons with previous malignancies effectively treated and not requiring treatment for >24 months are eligible, provided there is unambiguous documentation that current local recurrence or metastatic site represents recurrence of the primary breast malignancy.
  13. Patients who are HIV positive (by self-report) or have clinical or laboratory features indicative of AIDS.
  14. 14. Patients who require systemic steroids at a dose equivalent of >10 mg/day of prednisone. Beta-blocker therapy, while not exclusionary, is discouraged and alternatives should be sought if possible. The beta-blocker might compromise use of epinephrine for the rare possibility of anaphylaxis. Anticoagulants must be approved by the Investigator with notification of the Sponsor.
  15. Patients who are on treatment for rheumatological or autoimmune disease unless approved by the Investigator in consultation with the Sponsor (e.g., as for replacement therapy for autoimmune thyroiditis or diabetes).
  16. Patients with severe psychiatric (i.e. schizophrenia, bipolar, or borderline personality disorder) or other clinically progressive major medical problems, unless approved by the PI.
  17. Male breast cancer patients.
  18. Patients may not be on a concurrent clinical trial, unless approved by PI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, FACS, Study Director — Cancer Insight, LLC
Locations (5):
- United States (5):
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - University of Miami/Sylvester at Plantation, Plantation, Florida
  - Cancer Center of Kansas (CCK), Wichita, Kansas
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Providence Regional Medical Center, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://briacell.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SV-BR-1-GM Monotherapy
Started | 24
Completed | 14
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: Patients with Advanced Breast Cancer
Arm/Group | SV-BR-1-GM Monotherapy
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events Occurring in Two or More Patients [Safety]
Description: To evaluate the number of patients with toxicity events while on SV-BR-1-GM, as defined by the Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: Through study completion, an average of 1 year
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | SV-BR-1-GM Monotherapy
Number analyzed (Participants) | 24
Participants
  Patients with Adverse Events | 24
  Erythema injection site | 11
  Pruritis injection site | 8
  Induration injection site | 7
  Fatigue | 6
  Nausea | 6
  Constipation | 5
  Abdominal pain | 4
  Flu like symptoms | 4
  Diarrhea | 3
  GGTP increased | 3
  Injection site reaction | 3
  Urinary Tract Infection | 3
  Vomiting | 3
  Abdominal distension | 2
  Alkaline Phosphatase Increased | 2
  ALT Increased | 2
  Anorexia | 2
  AST Increased | 2
  Back Pain | 2
  Chills | 2
  Decreased appetite | 2
  Dehydration | 2
  Dizziness | 2
  Erythema Multiforme | 2
  Glucose increased | 2
  Hematocrit Decreased | 2
  Hypercalcemia | 2
  Lymphocytes Decreased | 2
  Myalgia | 2
  Pleural Effusion | 2

2. Secondary Outcome: Duration of Treatment Emergent Adverse Events [Safety]
Description: To evaluate the duration of toxicity events while on SV-BR-1-GM, as defined by CTCAE
Time Frame: Through study completion, an average of 1 year
Measure: Median (Full Range); unit: Days
Groups:
- Median Duration: Median duration of adverse events
Arm/Group | Median Duration
Number analyzed (Participants) | 24
Days | 8 [0 to 422]

3. Secondary Outcome: Number of Participants With an Adverse Event Related to SV-BR-1-GM Administration [Safety]
Description: To evaluate the number of participants with an adverse event related to SV-BR-1-GM administration, as defined by CTCAE
Time Frame: Through study completion, an average of 1 year
Population: Number with related adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | SV-BR-1-GM Monotherapy
Number analyzed (Participants) | 24
Participants | 23

4. Secondary Outcome: Objective Tumor Response Rate
Description: Objective response rate (ORR), defined as complete response (CR) or partial response (PR) per response evaluation criteria in solid tumors (RECIST) and immune-related RECIST (iRECIST) criteria.
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SV-BR-1-GM Monotherapy
Number analyzed (Participants) | 24
Participants | 0

5. Secondary Outcome: Rate of Non-progression of Tumors
Description: Non-progressive rate, defined as CR, PR or stable disease (SD) per RECIST and iRECIST criteria
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SV-BR-1-GM Monotherapy
Number analyzed (Participants) | 24
Participants | 4

6. Secondary Outcome: Durability of Tumor Response
Description: Durability of response, as defined as complete response (disappearance of all tumors), partial response (30% or greater reduction in the sum of diameters of target lesions (tumors) with stable disease in non-target lesions) or stable disease (less than 20% increase in the sum of diameters of target lesions with no new lesions appearing) by evaluating those patients eligible to complete the optional treatments from 9-12 months
Time Frame: Through study completion, an average of 1 year
Measure: Median (Full Range); unit: days
Arm/Group | SV-BR-1-GM Monotherapy
Number analyzed (Participants) | 24
days | 105.5 [79 to 197]

7. Other Pre Specified Outcome: Immune Responses to Vaccine
Description: To assess immune responses to SV-BR-1-GM, and to recall antigens, if any, as measured by DTH skin tests and/or other immunological tests
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Quality of Life Using the SF-36 Health Survey
Description: To measure the quality of life (QOL) of participants using the SF-36 Health Survey, which includes measures of General Health, Limitations of Activity, Physical Health Problems, Emotional Health Problems, Social Activities, Energy and Emotions.
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Weight
Description: To measure changes in weight.
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Performance Status
Description: To measure changes in performance status using the Eastern Cooperative Oncology Group (ECOG) scale
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Pain (Pain Scale)
Description: To measure changes in pain using a scale from None to Very Mild to Mild to Moderate to Severe to Very Severe
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: Used CTCAE V4.03 to determine adverse event intensity
Arm/Group | SV-BR-1-GM Monotherapy
All-Cause Mortality (participants affected / at risk) | 3/24
Serious Adverse Events (participants affected / at risk) | 8/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SV-BR-1-GM Monotherapy (N=24)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restrictive Cardiomyopathy (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Influenza A (Infections and infestations) | 1 (1)
Worsening of Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SV-BR-1-GM Monotherapy (N=24)
Erythema, injection site (General disorders) | 11 (42)
Pruritis, injection site (General disorders) | 8 (14)
Induration, injection site (General disorders) | 7 (31)
Fatigue (General disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 6 (8)
Constipation (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Flu like symptoms (General disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 3 (5)
GGTP increased (Investigations) | 3 (5)
Injection site reaction (General disorders) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Alkaline Phosphatase Increased (Investigations) | 2 (4)
ALT Increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
AST Increased (Investigations) | 2 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Glucose increased (Investigations) | 2 (2)
Hematocrit Decreased (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (4)
Lymphocytes Decreased (Investigations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
One patient dropped out after receiving cyclophosphamide and did not receive SV-BR-1-GM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03066947/Prot_SAP_000.pdf